CLINICAL TRIAL: NCT00399529
Title: A Feasibility Study of Combination Therapy With Trastuzumab, Cyclophosphamide, and an Allogeneic GM-CSF-secreting Breast Tumor Vaccine for HER-2/Neu-Overexpressing Metastatic Breast Cancer.
Brief Title: Trastuzumab, Cyclophosphamide, and an Allogeneic GM-CSF-secreting Breast Tumor Vaccine for the Treatment of HER-2/Neu-Overexpressing Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: American Cancer Society, Inc. (Other); Avon Foundation (Other); Cancer Treatment Research Foundation (Other); The Commonwealth Fund (Other); United States Department of Defense (U.S. Federal Agency); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J05118; RAC 0605-778; NCT00397371 (obsolete NCT alias)
Record Dates: First submitted 2006-11-13; First posted 2006-11-15 (Estimated); Results first posted 2020-04-13 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Breast Neoplasms
Keywords: Stage IV HER-2/neu overexpressing breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allo GM-CSF-secreting vaccine, Trastuzumab, Cyclophosphamide (Experimental): Allogeneic GM-CSF-secreting breast cancer vaccine : the vaccine containing a mixture of two GM-CSF-secreting allogeneic breast cancer cell lines (two parts 2T47D-V and one part 3SKBR3-7 mixed in a fixed dose of 5 X 10^8 cells for each patient and each vaccination cycle) given intradermally every 4-6 weeks for 3 cycles and then a 4th dose given 6-8 months after beginning the study.
  Trastuzumab : An initial loading dose of 4 mg/kg for participants beginning treatment with Trastuzumab, otherwise 2 mg/kg given every week intravenously
  Cyclophosphamide : 300 mg/m^2 given intravenously every 4-6 weeks for 3 cycles and then once 6-8 months after beginning the study
  Interventions: Biological: Allogeneic GM-CSF-secreting breast cancer vaccine; Drug: Trastuzumab; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Allogeneic GM-CSF-secreting breast cancer vaccine — the vaccine containing a mixture of two GM-CSF-secreting allogeneic breast cancer cell lines (two parts 2T47D-V and one part 3SKBR3-7 mixed in a fixed dose of 5 X 108 cells for each patient and each vaccination cycle) on day 0.
  Other Names: two parts 2T47D-V; one part 3SKBR3-7
Drug: Trastuzumab — Trastuzumab is a humanized monoclonal antibody specific for the extracellular domain of HER-2/neu that is now one component of the standard of care for both early and late stage HER-2/neu-overexpressing breast cancers. It exerts a pleiotropic antitumor effect by multiple mechanisms. The antibody decreases heterodimer formation with other members of the epidermal growth factor receptor (EGFR) family, thereby indirectly inhibiting signaling through the Ras/Raf/mitogen-activated protein kinases (MAPK) and Phosphatidylinositol 3-kinase(PI3K)/protein kinase B (Akt) pathways. It also inhibits tumor neovascularization, and augments apoptosis both in vitro and in vivo. Trastuzumab prevents cleavage of the extracellular domain of HER-2/neu, thus abrogating the constitutive activation of the remaining membrane-associated intracellular domain.
  Other Names: Herceptin
Drug: Cyclophosphamide — The doses of Cyclophosphamide are based on previously reported clinical experience as well as our own preclinical data demonstrating augmented vaccine efficacy with CY-modulated vaccination. In particular, 300 mg/m2
  Other Names: Cytoxan

SUMMARY:
This is a feasibility study to examine combination therapy with Trastuzumab (T), Cyclophosphamide (CY), and an allogeneic GM-CSF-secreting whole cell breast cancer vaccine in patients with Stage IV HER-2/neu-overexpressing breast cancer. The main purposes of this study are to test the safety, clinical benefit, and bioactivity of vaccine therapy in combination with Cyclophosphamide and Trastuzumab in patients with HER-2/neu-overexpressing Stage IV breast cancer. This study will also to test whether the Cyclophosphamide can eliminate the suppressive influence of regulatory T cells, and whether Trastuzumab can increase antigen processing and presentation. These drug activities may make the immune system react better and enhance the effects of the vaccine in treating breast cancer. The vaccine consists of two irradiated allogeneic mammary carcinoma cell lines genetically modified to secrete human granulocyte-macrophage colony stimulating factor (GM-CSF). This open label, single arm study is designed to recruit up to 40 subjects to identify 20 research subjects with HER-2/neu-overexpressing Stage IV breast cancer eligible for study treatment.

DETAILED DESCRIPTION:
Breast cancer ranks second among cancer deaths in women. In the year 2005, the American Cancer Society has estimated that 212,240 new invasive cases of breast cancer will be diagnosed, and predicts 40,410 deaths will result from breast cancer. While 80% of patients present with locoregional disease involving the breast and/or axillary lymph nodes, about half develop disseminated disease and ultimately die from it. Stage IV breast cancer is typically managed with hormonal agents or conventional cytotoxic drugs. Tumors quickly become resistant to these treatments. Immunotherapy is a particularly attractive strategy for overcoming drug resistance and can be integrated with existing therapeutic modalities in an additive or synergistic fashion. Immunotherapy is a type of treatment for cancer based on the idea that the immune system can be activated to destroy cancer cells that might be resistant to hormonal therapy and chemotherapy. A vaccine is a kind of immunotherapy that delivers an antigen (something that activates the immune system) so that the immune system recognizes cells with that antigen as foreign and destroys any cells that display that antigen.

The allogeneic breast tumor cell vaccine consists of two types of breast tumor cells developed from the tumor cells of patients with breast cancer. The human granulocyte-macrophage colony-stimulating factor (GM-CSF) gene was used to genetically modify the breast tumor cells to secrete GM-CSF. GM-CSF is a substance made by the body that helps the immune system recognize a tumor and destroy it. The vaccine cells were irradiated to prevent them from growing or dividing. The cells themselves are not radioactive. The cells are stored frozen until the day of vaccination. The total number of cells in each vaccine will be 500,000,000, divided into twelve injections given in the thighs and arms. The choice of twelve injections for each vaccine is based on the volume of the vaccine and a finding that the body has a better chance to respond to the vaccine if it is injected into a number of different areas.

We propose to test the safety and bioactivity of an allogeneic GM-CSF-secreting breast cancer vaccine when given in a specifically timed sequence with Cyclophosphamide and Trastuzumab, two drugs commonly used to treat breast cancer. In this study the Cyclophosphamide is used at lower doses than usual to help the vaccine to activate the patient's immune system. Trastuzumab will be given at doses that are commonly used to treat breast cancer and it may also increase the immune response. The dose and scheduling of Cyclophosphamide and Trastuzumab used are based on testing the drugs with a GM-CSF-secreting vaccine in mice that get breast cancer, and are the ones that enabled the vaccine to induce the most potent anti-tumor immunity. The dose of vaccine cells is based on the safety of the same dose of a similar GM-CSF-secreting vaccine for pancreatic cancer. This breast cancer vaccine has also been given to people with breast cancer by itself, and with Cyclophosphamide and another chemotherapy drug, Doxorubicin. To date, people have had no vaccine-related serious side effects, but not enough people have received the vaccine to know if it treats breast cancer. The vaccine is experimental and has not been approved by the U.S. Food and Drug Administration (FDA). However, the FDA has permitted its use in this research study. This is the second study of this breast cancer vaccine and the first study to test this vaccine with Trastuzumab.

The main purposes of this study are to test the safety, clinical benefit, and bioactivity of vaccine therapy in combination with Cyclophosphamide and Trastuzumab in patients with HER-2/neu-overexpressing Stage IV breast cancer. This study will also to test whether the Cyclophosphamide can eliminate the suppressive influence of regulatory T cells, and whether Trastuzumab can increase antigen processing and presentation. These drug activities may make the immune system react better and enhance the effects of the vaccine in treating breast cancer.

The study is open to men and women with HER-2/neu-overexpressing metastatic breast cancer. Concurrent hormone therapy and/or bisphosphonates (standard breast cancer therapy that is not chemotherapy or other investigational therapy) is allowed. Patients may have received Trastuzumab in the past or continue on it while participating in this study. About 40 people with HER-2/neu positive breast cancer will enter in the study. About 20 will pass the screening tests and receive the vaccine.

Research subjects will receive a fixed dose of the allogeneic breast tumor vaccine consisting of two irradiated allogeneic breast cancer cell lines transfected with the GM-CSF gene in a specifically timed sequence with a low dose of Cyclophosphamide and Trastuzumab. Patients will receive 300 mg/m2 of Cyclophosphamide on day -1, and the vaccine on day 0. Weekly Trastuzumab will be timed to coincide with Cyclophosphamide administration. Research subjects will receive three monthly vaccination cycles, with a fourth and final (boost) vaccination cycle three months from the third cycle.

Blood samples to measure GM-CSF levels will be taken on the day of vaccination, every day for 4 days, and then on day 7 after vaccination. Blood samples to evaluate the safety of the vaccinations will be taken about once a week for one month following each vaccination. During studies of the breast vaccine and similar vaccines in renal cell cancer, prostate cancer, pancreatic cancer, and non-small cell lung cancer, local symptoms of swelling and redness developed at the vaccine site between 2 and 7 days after vaccination. In this study, if the subject's vaccination site shows swelling over 1 cm in diameter, a skin biopsy will be taken. The skin biopsy will be evaluated to determine to what types of cells are important to the immune response. Based on our previous preclinical and clinical data, the biopsy will be taken on day 3, and possibly on day 7, after the first and third vaccinations. Other tests and evaluations include history and physical examination, vital signs, CT of the chest, abdomen, and pelvis, nuclear medicine bone scan, pre-vaccination biopsy, blood for immune monitoring, and a skin test for delayed-type hypersensitivity (DTH) that is like a purified protein derivative (PPD) test and involves injecting pieces of a protein antigen (HER-2/neu) that is delivered by the breast cancer vaccine. The purpose of the DTH test is to evaluate whether the research subject has developed a systemic immune response to the breast cancer vaccine. Tumor core needle biopsies will be obtained at baseline, and on days 0 and +14 of vaccine cycle 1 only.

Patients will be evaluated clinically and with laboratory testing for evidence of disease progression after each cycle or when otherwise clinically indicated. Computed tomography (CT scan) of the chest, abdomen, and pelvis and nuclear medicine bone scan will also be performed to evaluate disease status prior to starting the study, after vaccine cycle 3 and prior to and after vaccine cycle 4. About every three months cardiac function will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed HER-2/neu-overexpressing adenocarcinoma of the breast; this is defined as HER-2+ by immunohistochemistry (IHC) 3+ staining or Fluorescence In-Situ Hybridization (FISH). Prior adjuvant Trastuzumab therapy is permitted. Patients must not be eligible for therapy of known curative potential for metastatic breast cancer if it is identified during the course of the study.
2. Patients may have measurable or evaluable disease.
3. Stable central nervous system (CNS) disease that has been adequately treated and is not under active treatment allowed.
4. Age 18 years or older.
5. Able to give informed consent.
6. Patients with an Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1.
7. No systemic oral steroids administered within 28 days prior to initiating treatment on protocol. Topical, ocular, and nasal steroids are allowed, as are those applied to mucus membranes.
8. No prior or currently active autoimmune disease requiring management with systemic immunosuppression. This includes inflammatory bowel disease, systemic vasculitis, scleroderma, psoriasis, multiple sclerosis, hemolytic anemia or immune-mediated thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjogren's syndrome, sarcoidosis, or other rheumatologic disease. Asthma or chronic obstructive pulmonary disease that does not require daily systemic corticosteroids is acceptable.
9. Not pregnant, and on appropriate birth control if of child-bearing potential.
10. No history of other malignancies within the prior five years (excluding a history of carcinoma in situ of the cervix, superficial non-melanoma skin cancer, and superficial bladder cancer).
11. Adequate bone marrow reserve with absolute neutrophil count (ANC) > 1000 and platelets > 100,000.
12. Adequate renal function with serum creatinine < 2.0.
13. Adequate hepatic reserve with serum bilirubin < 2.0, aspartate transaminase (AST) and alanine aminotransferase (ALT) < 2X the upper limit of normal, and alkaline phosphatase < 5X the upper limit of normal. Serum bilirubin > 2.0 is acceptable in the setting of known Gilbert's syndrome.
14. Adequate cardiac reserve with a cardiac ejection fraction within the lower limit of facility normal by MUGA, or 45% by echocardiogram.
15. No active major medical or psychosocial problems that could be complicated by study participation.
16. HIV negative.

Exclusion Criteria:

1. No histologic documentation of breast adenocarcinoma.
2. Breast adenocarcinoma that is not amplified for HER-2/neu gene expression by at least 2-fold by FISH analysis, or that is less than IHC 3+ when FISH negative.
3. Cardiac dysfunction documented by an ejection fraction less than the lower limit of the facility normal by multi-gated acquisition (MUGA) scan, or 45% by echocardiogram.
4. Symptomatic intrinsic lung disease or extensive tumor involvement of the lungs resulting in dyspnea at rest.
5. History of autoimmune disease as detailed above.
6. Systemic oral corticosteroid treatment within 28 days prior to initiating treatment on study.
7. Uncontrolled medical problems.
8. Evidence of active acute or chronic infection.
9. Chemotherapy, radiation therapy, or biologic therapy (except Trastuzumab) within 28 days prior to initiating treatment on study. Hormonal therapy and supportive therapy with bisphosphonates will be allowed.
10. Participation in an investigational new drug trial within 28 days prior to initiating treatment on study.
11. Pregnant or breast feeding.
12. Hepatic, renal, or bone marrow dysfunction as detailed above.
13. Concurrent malignancy or history of other malignancy within the last five years except as noted above.
14. Corn allergy.
15. Known severe hypersensitivity to Trastuzumab (excluding mild to moderate infusion reactions that are easily managed and do not recur).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leisha A Emens, M.D.,Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Chen G, Gupta R, Petrik S, Laiko M, Leatherman JM, Asquith JM, Daphtary MM, Garrett-Mayer E, Davidson NE, Hirt K, Berg M, Uram JN, Dauses T, Fetting J, Duus EM, Atay-Rosenthal S, Ye X, Wolff AC, Stearns V, Jaffee EM, Emens LA. A feasibility study of cyclophosphamide, trastuzumab, and an allogeneic GM-CSF-secreting breast tumor vaccine for HER2+ metastatic breast cancer. Cancer Immunol Res. 2014 Oct;2(10):949-61. doi: 10.1158/2326-6066.CIR-14-0058. Epub 2014 Aug 12. PMID 25116755

RESULTS

PARTICIPANT FLOW:
Groups:
- Allo GM-CSF-secreting Vaccine, Trastuzumab, Cyclophosphamide: Allogeneic granulocyte-macrophage colony-stimulating factor (GM-CSF)-secreting breast cancer vaccine: the vaccine containing a mixture of two GM-CSF-secreting allogeneic breast cancer cell lines (two parts 2T47D-V and one part 3SKBR3-7 mixed in a fixed dose of 5 X 10^8 cells for each patient and each vaccination cycle) given intradermally every 4-6 weeks for 3 cycles and then a 4th dose given 6-8 months after beginning the study.
  Cyclophosphamide (Cy): 300 mg/m^2 given intravenously every 4-6 weeks for 3 cycles and then once 6-8 months after beginning the study
  Trastuzumab : An initial loading dose of 4 mg/kg for participants beginning treatment with Trastuzumab, otherwise 2 mg/kg given every week intravenously
Period: Overall Study
Arm/Group | Allo GM-CSF-secreting Vaccine, Trastuzumab, Cyclophosphamide
Started | 22
Completed | 20
Not Completed | 2
Not completed — Off Study Prior to Treatment | 2

BASELINE CHARACTERISTICS:
Groups:
- Allo GM-CSF-secreting Vaccine, Trastuzumab, Cyclophosphamide: Allogeneic GM-CSF-secreting breast cancer vaccine : the vaccine containing a mixture of two GM-CSF-secreting allogeneic breast cancer cell lines (two parts 2T47D-V and one part 3SKBR3-7 mixed in a fixed dose of 5 X 10^8 cells for each patient and each vaccination cycle) given intradermally every 4-6 weeks for 3 cycles and then a 4th dose given 6-8 months after beginning the study.
  Cyclophosphamide : 300 mg/m^2 given intravenously every 4-6 weeks for 3 cycles and then once 6-8 months after beginning the study
  Trastuzumab : An initial loading dose of 4 mg/kg for participants beginning treatment with Trastuzumab, otherwise 2 mg/kg given every week intravenously
Arm/Group | Allo GM-CSF-secreting Vaccine, Trastuzumab, Cyclophosphamide
Number analyzed (Participants) | 22
Age, Continuous [Mean (Full Range); unit: years] | 52 [34 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Safety is measured as the number of patients that experienced adverse events related to study drug.
Time Frame: From first dose through 30 days after last dose of study drug, up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Allo GM-CSF-secreting Vaccine, Trastuzumab, Cyclophosphamide
Number analyzed (Participants) | 20
Participants
  Fatigue | 8
  Urticaria | 7
  Pruritus | 6
  Fever | 5
  Flu-like symptoms | 4
  Lymphadenopathy | 4
  Abdominal pain | 3
  Rash | 3
  Malaise | 3
  Chills | 3
  Dizziness | 2
  Anorexia | 1
  Erythema | 1
  Headache | 1
  Nausea | 1
  Arm pain | 1
  Cancer site pain | 1
  Leg pain | 1
  Groin tightness | 1
  Erythema at vaccine sites | 20
  Pruritus at vaccine sites | 20
  Induration at vaccine sites | 20
  Pain at vaccine sties | 17
  Rash at vaccine sites | 7
  Blister at vaccine sites | 5
  Hyperpigmentation at vaccine sites | 4
  Bruising at vaccine sites | 3
  Edema at vaccine sites | 2
  Vaccine site flare | 2

2. Primary Outcome: Number of Participants With Clinical Benefit
Description: Clinical benefit is defined as the proportion of patients achieving complete response, partial response, or stable disease by RECIST. Complete response (CR) is defined as total disappearance of all clinical evidence of reversible disease. A partial response (PR) is defined as a >=30% reduction in tumor target lesions. Stable disease (SD) is defined as disease status that fails to qualify as as a response (CR or PR) or progressive disease (increase of at least 20% in tumor target lesions).
Time Frame: At 6 and 12 months from start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Allo GM-CSF-secreting Vaccine, Trastuzumab, Cyclophosphamide
Number analyzed (Participants) | 20
Participants
  Clinical Benefit at 6 months | 11
  Clinical Benefit at 12 months | 8

3. Secondary Outcome: Number of Participants With Delayed Type Hypersensitivity (Immunological Response)
Description: The number of participants with a Delayed Type Hypersensitivity (DTH) response was measured as an indicator of immune response. Participants were considered to have a DTH response if they had increased induration (>5mm from baseline) at the site of injection 2-3 days after intradermal injection with human epidermal growth factor receptor 2 (HER-2) peptides. This peptide injection was given 28 days after each dose of vaccine.
Time Frame: 30 days after each vaccine, up to 9 months
Measure: Count of Participants; unit: Participants
Groups:
- Allo GM-CSF-secreting Vaccine, Trastuzumab, Cyclophosphamide: Allogeneic GM-CSF-secreting breast cancer vaccine :
  5 X 10^8 cells given intradermally every 4-6 weeks for 3 cycles and then a 4th dose given 6-8 months after beginning the study.
  Cyclophosphamide : 300 mg/m^2 given intravenously every 4-6 weeks for 3 cycles and then once 6-8 months after beginning the study
  Trastuzumab : An initial loading dose of 4 mg/kg for participants beginning treatment with Trastuzumab, otherwise 2 mg/kg given every week intravenously
Arm/Group | Allo GM-CSF-secreting Vaccine, Trastuzumab, Cyclophosphamide
Number analyzed (Participants) | 20
Participants | 7

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from first dose through 30 days after last dose of study drugs, up to 9 months.
Arm/Group | Allo GM-CSF-secreting Vaccine, Trastuzumab, Cyclophosphamide
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Allo GM-CSF-secreting Vaccine, Trastuzumab, Cyclophosphamide (N=20)
Urticaria (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Allo GM-CSF-secreting Vaccine, Trastuzumab, Cyclophosphamide (N=20)
Fatigue (General disorders) | 8
Urticaria (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 6
Fever (General disorders) | 5
Flu-like symptoms (General disorders) | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 4
Abdominal Pain (Gastrointestinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Malaise (General disorders) | 3
Chills (General disorders) | 3
Dizziness (Nervous system disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Headache (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Arm Pain (Musculoskeletal and connective tissue disorders) | 1
Cancer Site Pain (General disorders) | 1
Leg Pain (Musculoskeletal and connective tissue disorders) | 1
Erythema at Vaccine Sites (General disorders) | 20
Pruritus at Vaccine Sites (General disorders) | 20
Pain at Vaccine Sites (General disorders) | 17
Rash at Vaccine Sites (General disorders) | 7
Blister at Vaccine Sites (General disorders) | 5
Hyperpigmentation at Vaccine Sites (General disorders) | 4
Bruising at Vaccine Sites (General disorders) | 3
Edema at Vaccine Sites (General disorders) | 2
Vaccine Site Flares (General disorders) | 2
Groin Tightness (Musculoskeletal and connective tissue disorders) | 1
Induration at Vaccine Sites (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No